CLINICAL TRIAL: NCT06133816
Title: Using a Simplified Tool to Predict Lung Cancer Screening (LCS) Eligibility: Experiment to Test Effects of Messaging on Response Rates
Brief Title: Lung Cancer Screening Eligibility Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katharine Rendle, Assistant Professor, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: UPCC 16523; P50CA271338-02 (NIH); 853337 (Other: UPenn IRB)
Record Dates: First submitted 2023-10-18; First posted 2023-11-18 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: We will use a randomized factorial design to test the effects of different types of messaging with or without incentives on response rates to an eligibility survey.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Arm 1 (Introductory Message A + Tobacco Use Message A + Incentive) (Experimental): Participants will receive two framed messages (AA) plus an incentive
  Interventions: Behavioral: Framed Introductory Message A; Behavioral: Framed Tobacco Use Message A; Behavioral: Financial Incentive
- Arm 2 (Introductory Message A + Tobacco Use Message A) (Experimental): Participants will receive two framed messages (AA)
  Interventions: Behavioral: Framed Introductory Message A; Behavioral: Framed Tobacco Use Message A
- Arm 3 (Introductory Message A + Tobacco Use Message B + Incentive) (Experimental): Participants will receive two framed messages (AB) plus an incentive
  Interventions: Behavioral: Framed Introductory Message A; Behavioral: Framed Tobacco Use Message B; Behavioral: Financial Incentive
- Arm 4 (Introductory Message A + Tobacco Use Message B) (Experimental): Participants will receive two framed messages (AB)
  Interventions: Behavioral: Framed Introductory Message A; Behavioral: Framed Tobacco Use Message B
- Arm 5 (Introductory Message B + Tobacco Use Message A + Incentive) (Experimental): Participants will receive two framed messages (BA) plus an incentive
  Interventions: Behavioral: Framed Introductory Message B; Behavioral: Framed Tobacco Use Message A; Behavioral: Financial Incentive
- Arm 6 (Introductory Message B + Tobacco Use Message A) (Experimental): Participants will receive two framed messages (BA)
  Interventions: Behavioral: Framed Introductory Message B; Behavioral: Framed Tobacco Use Message A
- Arm 7 (Introductory Message B + Tobacco Use Message B + Incentive) (Experimental): Participants will receive two framed messages (BB) plus an incentive
  Interventions: Behavioral: Framed Introductory Message B; Behavioral: Framed Tobacco Use Message B; Behavioral: Financial Incentive
- Arm 8 (Introductory Message B + Tobacco Use Message B) (Experimental): Participants will receive two framed messages (BB)
  Interventions: Behavioral: Framed Introductory Message B; Behavioral: Framed Tobacco Use Message B
- Arm 9 (Introductory Message C + Tobacco Use Message A + Incentive) (Experimental): Participants will receive two framed messages (CA) plus an incentive
  Interventions: Behavioral: Framed Introductory Message C; Behavioral: Framed Tobacco Use Message A; Behavioral: Financial Incentive
- Arm 10 (Introductory Message C + Tobacco Use Message A) (Experimental): Participants will receive two framed message (CA)
  Interventions: Behavioral: Framed Introductory Message C; Behavioral: Framed Tobacco Use Message A
- Arm 11 (Introductory Message C + Tobacco Use Message B + Incentive) (Experimental): Participants will receive two framed messages (CB) plus an incentive
  Interventions: Behavioral: Framed Introductory Message C; Behavioral: Framed Tobacco Use Message B; Behavioral: Financial Incentive
- Arm 12 (Introductory Message C + Tobacco Use Message B) (Experimental): Participants will receive two framed messages (CB)
  Interventions: Behavioral: Framed Introductory Message C; Behavioral: Framed Tobacco Use Message B

INTERVENTIONS:
Behavioral: Framed Introductory Message A — Randomly assign patients to receive introductory message encouraging them to complete the survey (version A).
  Arms: Arm 1 (Introductory Message A + Tobacco Use Message A + Incentive); Arm 2 (Introductory Message A + Tobacco Use Message A); Arm 3 (Introductory Message A + Tobacco Use Message B + Incentive); Arm 4 (Introductory Message A + Tobacco Use Message B)
Behavioral: Framed Introductory Message B — Randomly assign patients to receive introductory message encouraging them to complete the survey (version B).
  Arms: Arm 5 (Introductory Message B + Tobacco Use Message A + Incentive); Arm 6 (Introductory Message B + Tobacco Use Message A); Arm 7 (Introductory Message B + Tobacco Use Message B + Incentive); Arm 8 (Introductory Message B + Tobacco Use Message B)
Behavioral: Framed Introductory Message C — Randomly assign patients to receive introductory message encouraging them to complete the survey (version C).
  Arms: Arm 10 (Introductory Message C + Tobacco Use Message A); Arm 11 (Introductory Message C + Tobacco Use Message B + Incentive); Arm 12 (Introductory Message C + Tobacco Use Message B); Arm 9 (Introductory Message C + Tobacco Use Message A + Incentive)
Behavioral: Framed Tobacco Use Message A — Randomly assign patients to receive norming message related to tobacco use (version A).
  Arms: Arm 1 (Introductory Message A + Tobacco Use Message A + Incentive); Arm 10 (Introductory Message C + Tobacco Use Message A); Arm 2 (Introductory Message A + Tobacco Use Message A); Arm 5 (Introductory Message B + Tobacco Use Message A + Incentive); Arm 6 (Introductory Message B + Tobacco Use Message A); Arm 9 (Introductory Message C + Tobacco Use Message A + Incentive)
Behavioral: Framed Tobacco Use Message B — Randomly assign patients to receive norming message related to tobacco use (version B).
  Arms: Arm 11 (Introductory Message C + Tobacco Use Message B + Incentive); Arm 12 (Introductory Message C + Tobacco Use Message B); Arm 3 (Introductory Message A + Tobacco Use Message B + Incentive); Arm 4 (Introductory Message A + Tobacco Use Message B); Arm 7 (Introductory Message B + Tobacco Use Message B + Incentive); Arm 8 (Introductory Message B + Tobacco Use Message B)
Behavioral: Financial Incentive — Randomly assigned patients to be entered into a drawing to receive a $100 gift card.
  Arms: Arm 1 (Introductory Message A + Tobacco Use Message A + Incentive); Arm 11 (Introductory Message C + Tobacco Use Message B + Incentive); Arm 3 (Introductory Message A + Tobacco Use Message B + Incentive); Arm 5 (Introductory Message B + Tobacco Use Message A + Incentive); Arm 7 (Introductory Message B + Tobacco Use Message B + Incentive); Arm 9 (Introductory Message C + Tobacco Use Message A + Incentive)

SUMMARY:
The primary purpose of this study evaluate if different messaging impacts response rates to a brief survey (i.e., the simplified eligibility tool) that is designed to estimate pack-year eligibility for lung cancer screening (LCS). This will help inform the best way to increase response rates to the tool in future intervention studies designed to increase LCS, and expand upon survey methodology in general.

DETAILED DESCRIPTION:
Despite growing evidence that lung cancer screening (LCS) reduces lung cancer-specific mortality, LCS across the United States is remarkably low. This is due in part to challenges with identifying adults who meet eligibility criteria for lifetime smoking intensity (i.e., 20 pack-years or greater), which is often missing from the electronic medical record. We have developed a simplified eligibility tool that has shown accuracy in estimating pack-years. But given the potential for low response rates, there is a great need to identify effective strategies to increasing response rates equitably prior to using it in practice or in future studies. The primary purpose of this study evaluate if different messaging impacts response rates to a brief survey (i.e., the simplified eligibility tool) that is designed to estimate pack-year eligibility for lung cancer screening (LCS). This will help to identify the best way to increase response rates to the tool in future intervention studies designed to increase LCS, and expand upon survey methodology in general.

ELIGIBILITY:
Inclusion Criteria:

1. meet age eligibility (50-80 years old) for LCS based on 2021 USPSTF guidelines; and
2. have completed at least one primary care visit at Penn Medicine in 2020-2025

Exclusion Criteria:

1. have a documented history of lung cancer;
2. have a documented history of completing LCS at Penn Medicine;
3. are listed as not wanting to be contacted or solicited for research; or
4. do not otherwise meet inclusion criteria.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6125 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine A Rendle, PhD,MSW,MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events
Period: Overall Study
Arm/Group | Arm 1 (Introductory Message A + Tobacco Use Message A + Incentive) | Arm 2 (Introductory Message A + Tobacco Use Message A) | Arm 3 (Introductory Message A + Tobacco Use Message B + Incentive) | Arm 4 (Introductory Message A + Tobacco Use Message B) | Arm 5 (Introductory Message B + Tobacco Use Message A + Incentive) | Arm 6 (Introductory Message B + Tobacco Use Message A) | Arm 7 (Introductory Message B + Tobacco Use Message B + Incentive) | Arm 8 (Introductory Message B + Tobacco Use Message B) | Arm 9 (Introductory Message C + Tobacco Use Message A + Incentive) | Arm 10 (Introductory Message C + Tobacco Use Message A) | Arm 11 (Introductory Message C + Tobacco Use Message B + Incentive) | Arm 12 (Introductory Message C + Tobacco Use Message B)
Started | 509 | 509 | 515 | 509 | 510 | 510 | 512 | 509 | 511 | 511 | 509 | 511
Completed | 509 | 509 | 515 | 509 | 510 | 510 | 512 | 509 | 511 | 511 | 509 | 511
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Introductory Message A + Tobacco Use Message A + Incentive) | Arm 2 (Introductory Message A + Tobacco Use Message A) | Arm 3 (Introductory Message A + Tobacco Use Message B + Incentive) | Arm 4 (Introductory Message A + Tobacco Use Message B) | Arm 5 (Introductory Message B + Tobacco Use Message A + Incentive) | Arm 6 (Introductory Message B + Tobacco Use Message A) | Arm 7 (Introductory Message B + Tobacco Use Message B + Incentive) | Arm 8 (Introductory Message B + Tobacco Use Message B) | Arm 9 (Introductory Message C + Tobacco Use Message A + Incentive) | Arm 10 (Introductory Message C + Tobacco Use Message A) | Arm 11 (Introductory Message C + Tobacco Use Message B + Incentive) | Arm 12 (Introductory Message C + Tobacco Use Message B) | Total
Number analyzed (Participants) | 509 | 509 | 515 | 509 | 510 | 510 | 512 | 509 | 511 | 511 | 509 | 511 | 6125
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.02 (0.35) | 64.33 (0.33) | 64.50 (0.33) | 64.48 (0.34) | 64.15 (0.33) | 64.67 (0.34) | 64.21 (0.33) | 63.33 (0.35) | 64.56 (0.33) | 64.28 (0.36) | 64.40 (0.33) | 63.89 (0.32) | 64.32 (0.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 260 | 261 | 258 | 259 | 259 | 261 | 258 | 260 | 259 | 258 | 260 | 3112
  Male | 250 | 249 | 254 | 251 | 251 | 251 | 251 | 251 | 251 | 252 | 251 | 251 | 3013
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 14 | 15 | 11 | 16 | 10 | 8 | 15 | 16 | 9 | 9 | 6 | 136
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 502 | 495 | 500 | 498 | 494 | 500 | 504 | 494 | 495 | 502 | 500 | 505 | 5989
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 0 | 2 | 2 | 0 | 1 | 1 | 4 | 3 | 4 | 21
  Asian | 6 | 6 | 6 | 12 | 8 | 8 | 10 | 8 | 5 | 7 | 14 | 7 | 97
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Black or African American | 94 | 94 | 95 | 93 | 95 | 95 | 95 | 94 | 94 | 94 | 94 | 94 | 1131
  White | 369 | 372 | 365 | 360 | 361 | 362 | 367 | 358 | 363 | 369 | 359 | 353 | 4358
  More than one race | 12 | 13 | 10 | 11 | 11 | 12 | 13 | 14 | 15 | 9 | 13 | 14 | 147
  Unknown or Not Reported | 26 | 23 | 37 | 33 | 32 | 31 | 27 | 34 | 32 | 28 | 26 | 39 | 368

OUTCOME MEASURES:

1. Primary Outcome: Full Survey Completion
Description: The proportion of participants that answers all three survey questions via text message among all those randomized.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Introductory Message A + Tobacco Use Message A + Incentive) | Arm 2 (Introductory Message A + Tobacco Use Message A) | Arm 3 (Introductory Message A + Tobacco Use Message B + Incentive) | Arm 4 (Introductory Message A + Tobacco Use Message B) | Arm 5 (Introductory Message B + Tobacco Use Message A + Incentive) | Arm 6 (Introductory Message B + Tobacco Use Message A) | Arm 7 (Introductory Message B + Tobacco Use Message B + Incentive) | Arm 8 (Introductory Message B + Tobacco Use Message B) | Arm 9 (Introductory Message C + Tobacco Use Message A + Incentive) | Arm 10 (Introductory Message C + Tobacco Use Message A) | Arm 11 (Introductory Message C + Tobacco Use Message B + Incentive) | Arm 12 (Introductory Message C + Tobacco Use Message B)
Number analyzed (Participants) | 509 | 509 | 515 | 509 | 510 | 510 | 512 | 509 | 511 | 511 | 509 | 511
Participants | 358 | 381 | 383 | 389 | 372 | 399 | 386 | 402 | 335 | 397 | 373 | 366

2. Secondary Outcome: Partial Survey Completion
Description: The proportion of participants that answer at least one of three survey questions via text message among all those randomized.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Introductory Message A + Tobacco Use Message A + Incentive) | Arm 2 (Introductory Message A + Tobacco Use Message A) | Arm 3 (Introductory Message A + Tobacco Use Message B + Incentive) | Arm 4 (Introductory Message A + Tobacco Use Message B) | Arm 5 (Introductory Message B + Tobacco Use Message A + Incentive) | Arm 6 (Introductory Message B + Tobacco Use Message A) | Arm 7 (Introductory Message B + Tobacco Use Message B + Incentive) | Arm 8 (Introductory Message B + Tobacco Use Message B) | Arm 9 (Introductory Message C + Tobacco Use Message A + Incentive) | Arm 10 (Introductory Message C + Tobacco Use Message A) | Arm 11 (Introductory Message C + Tobacco Use Message B + Incentive) | Arm 12 (Introductory Message C + Tobacco Use Message B)
Number analyzed (Participants) | 509 | 509 | 515 | 509 | 510 | 510 | 512 | 509 | 511 | 511 | 509 | 511
Participants | 377 | 405 | 394 | 403 | 381 | 414 | 403 | 408 | 345 | 413 | 383 | 385

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during active trial participation defined as days between randomization and end of participation (no more than 7 days).
Arm/Group | Arm 1 (Introductory Message A + Tobacco Use Message A + Incentive) | Arm 2 (Introductory Message A + Tobacco Use Message A) | Arm 3 (Introductory Message A + Tobacco Use Message B + Incentive) | Arm 4 (Introductory Message A + Tobacco Use Message B) | Arm 5 (Introductory Message B + Tobacco Use Message A + Incentive) | Arm 6 (Introductory Message B + Tobacco Use Message A) | Arm 7 (Introductory Message B + Tobacco Use Message B + Incentive) | Arm 8 (Introductory Message B + Tobacco Use Message B) | Arm 9 (Introductory Message C + Tobacco Use Message A + Incentive) | Arm 10 (Introductory Message C + Tobacco Use Message A) | Arm 11 (Introductory Message C + Tobacco Use Message B + Incentive) | Arm 12 (Introductory Message C + Tobacco Use Message B)
All-Cause Mortality (participants affected / at risk) | 0/509 | 0/509 | 0/515 | 0/509 | 0/510 | 0/510 | 0/512 | 0/509 | 0/511 | 0/511 | 0/509 | 0/511
Serious Adverse Events (participants affected / at risk) | 0/509 | 0/509 | 0/515 | 0/509 | 0/510 | 0/510 | 0/512 | 0/509 | 0/511 | 0/511 | 0/509 | 0/511
Other Adverse Events (participants affected / at risk) | 0/509 | 0/509 | 0/515 | 0/509 | 0/510 | 0/510 | 0/512 | 0/509 | 0/511 | 0/511 | 0/509 | 0/511

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT06133816/Prot_001.pdf
  • Statistical Analysis Plan (2023-11-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT06133816/SAP_000.pdf